CLINICAL TRIAL: NCT00990496
Title: A Phase I-II Study of Allogeneic CMV Specific Cytotoxic T Lymphocytes (CTL) for Patients With Refractory Glioblastoma Multiforme (GBM)
Brief Title: A Study Using Allogenic-Cytomegalovirus (CMV) Specific Cells for Glioblastoma Multiforme (GBM)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual goals not met
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31717; PSHCI #09-045
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma multiforme; GBM; Cytomegalovirus; CMV; Cytotoxic T lymphocyte; CTL
MeSH Terms: conditions — Glioblastoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GBM Treatment (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CMV Specific Cytotoxic T Lymphocytes (CTL)

INTERVENTIONS:
Drug: Fludarabine — 30 mg/m2
Drug: Cyclophosphamide — 600 mg/m2
Biological: CMV Specific Cytotoxic T Lymphocytes (CTL) — CTL Infusion (3 - 5 x 10E6 cells/kg)

SUMMARY:
The primary purpose of this study is to determine the safety and efficacy of the infusion of partially matched, allogeneic, CMV specific cytotoxic T cells (CTL) for patients with GBM that have failed primary therapy.

DETAILED DESCRIPTION:
Tumor specimens of consenting patients will be tested by immunohistochemistry (IHC) for the presence of IE-1 and/or pp65. Subjects whose tumors test positive for either or both CMV antigens will be consented for the treatment phase which will include a regimen of fludarabine and cyclophosphamide daily for two days, cyclophosphamide only for a third day, followed by one day of rest prior to the day of CTL infusion.

This trial intended to be a Phase 1/2 trial, but it never progressed to Phase 2 before termination.

ELIGIBILITY:
Inclusion Criteria:

FOR SCREENING

* Patients must have a histopathologic diagnosis of GBM.
* Patients from 5 to 65 years of age with GBM.

FOR TREATMENT

* GBM has progressed following primary therapy.
* Tumor is CMV pp65 or IE1 positive by immunohistochemistry (IHC).
* Subjects must have pulse oximetry > or = 94 % on no supplemental oxygen.
* Creatinine clearance must be > 50 cc/min as estimated by patient's serum creatinine, weight, and age.
* Bilirubin must be < 2.0 mg/dl and SGOT/SGPT < 2.5 X normal.
* ECOG performance status must be < or = 2, and for patients <16 years of age, Lansky performance status must be > or = 70%.

Exclusion Criteria:

* Pregnant females
* Subjects who are moribund or who because of cardiac, pulmonary, renal, hepatic or neurologic dysfunction are not expected to survive one month following the T cell infusion

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2010-10-28 (Actual); Study Completion 2010-10-28 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of tumor responses, as defined as stable disease, partial, or complete responses after the infusion of CMV CTL. | 2 years

SECONDARY OUTCOMES:
To determine the duration and magnitude of donor chimerism post infusion by micro chimerism assays. | 2 years
To determine the incidence of increases in CMV pp65 or IE-1 T cells post infusion of allogeneic CMV CTL of GBM patients. | 2 years
To determine safety of allogeneic CTL infusions in this patient population. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lucas G. Lucas, MD, Study Chair — Milton S. Hershey Medical Center